CLINICAL TRIAL: NCT05390853
Title: Pilot Randomized Controlled Study on Neuromodulation Through Active tDCS Versus Sham tDCS to Support Upper Limb Motor and Functional Recovery in Sub-acute, Incomplete, Tetraplegic Spinal Cord Injured Patients
Brief Title: Active tDCS Versus Sham tDCS for Upper Limb Recovery in Incomplete Tetraplegic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE AVEC_96-2022-SPER-AUSLIM
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Neuromodulation; Transcranial Direct Current Stimulation; tDCS; Upper limb; Functional recovery; Early rehabilitation; Incomplete tetraplegia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After selection, enrollment and basal assessments, patients are randomized just before the first tDCS session by the professional who will apply the tDCS and will thus be the only one knowing the assigned intervention during the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (A) (Experimental): Two daily tDCS sessions for 5 days a week, for 2 consecutive weeks, are carried out, simultaneously with the usual rehabilitation physiotherapy of the upper limbs.
  Patients will receive the usual rehabilitation physiotherapy of the upper limbs at least in the 4 weeks before and in the 4 weeks after the tDCS treatment period too.
  Interventions: Procedure: Active tDCS
- Sham tDCS (S) (Placebo Comparator): Two daily tDCS sessions for 5 days a week, for 2 consecutive weeks, are carried out, simultaneously with the usual rehabilitation physiotherapy of the upper limbs.
  Patients will receive the usual rehabilitation physiotherapy of the upper limbs at least in the 4 weeks before and in the 4 weeks after the tDCS treatment period too.
  Interventions: Procedure: Sham tDCS

INTERVENTIONS:
Procedure: Active tDCS — tDCS application is anodic, in the M1 area (Primary Motor Cortex) right or left, contralateral to the pre-defined target limb. The cathode is positioned in the supraorbital area, contralateral to the anode.
  Active stimulation is carried out with a current intensity of 2 milliAmpere. Each tDCS session lasts 20 minutes. tDCS is administered simultaneously during the first 20 minutes of the usual upper limb rehabilitation physiotherapy, which will continue for a further 20 minutes.
  During the whole study period (10 weeks) each patient is not subjected to any focal treatments in the target upper limb.
  In the study period, the contralateral limb is rehabilitated and evaluated according to usual practice.
  Arms: Active tDCS (A)
Procedure: Sham tDCS — tDCS application is anodic, in the M1 area (Primary Motor Cortex) right or left, contralateral to the pre-defined target limb. The cathode is positioned in the supraorbital area, contralateral to the anode.
  Sham stimulation is carried out through a dedicated program, which increases the current for several seconds up to the target intensity and then decreases it gradually in a few seconds, so that subjects experience the same itching and tingling experience as in active stimulation, but they do not receive any significant therapeutic currents.
  Each tDCS session lasts 20 minutes. tDCS is administered simultaneously during the first 20 minutes of the usual upper limb rehabilitation physiotherapy, which will continue for a further 20 minutes.
  During the whole study period (10 weeks) each patient is not subjected to any focal treatments in the target upper limb.
  In the study period, the contralateral limb is rehabilitated and evaluated according to usual practice.
  Arms: Sham tDCS (S)

SUMMARY:
Spinal Cord Injury (SCI) at the cervical level results in motor and sensory impairment below the lesion level and may determine a consistent loss of the use of the upper limbs, with a substantial impact on daily life activities. Therefore, functionality recovery of the upper limbs, of the hands in particular, represents a priority rehabilitation target. Studies in the literature show that the most relevant recovery occurs in the first months after SCI and that neuromodulation techniques may facilitate it. Transcranial Direct Current Stimulation (tDCS ) is a non-invasive neuromodulation technique. The present pilot, randomized controlled study aims at exploring the feasibility and efficacy of an early application of tDCS, in addition to the traditional physiotherapy treatment for the functional recovery of the upper limb, in incomplete traumatic tetraplegic subjects in the sub-acute phase after SCI occurrence. Patients hospitalized at the Montecatone Rehabilitation Institute are randomly assigned to Active tDCS or Sham tDCS.

DETAILED DESCRIPTION:
Spinal Cord Injury (SCI) at the cervical level results in motor and sensory impairment below the lesion level and may determine a consistent loss of the use of the upper limbs, with a substantial impact on daily life activities. Therefore, functionality recovery of upper limbs, of the hands in particular, represents a priority rehabilitation target. In cases of incomplete tetraplegia, the main rehabilitation goal is the recovery of the maximum functional capacity, in order to improve autonomy or, in the most serious cases, avoid complications due to immobilization.

Studies in the literature show that the most relevant recovery occurs in the first months after SCI and that neuromodulation techniques may facilitate it.

Transcranial Direct Current Stimulation (tDCS ) is a non-invasive neuromodulation technique capable of modifying cortical excitability through direct, low intensity current, generated by a programmable medical device and delivered through electrodes placed on the scalp. Some authors have explored its potential role in facilitating functional recovery and treating spasticity in SCI subjects, however there are few studies on the use of neuromodulation induced by tDCS as an aid for the functional recovery of upper limbs in tetraplegic subjects. Moreover, most of such studies are on chronic SCI persons only.

The present pilot, randomized controlled study aims at exploring the feasibility and efficacy of an early application of tDCS, in the sub-acute phase after SCI occurrence, for the functional recovery of the upper limb, in addition to the traditional physiotherapy treatment, in incomplete traumatic tetraplegic patients, hospitalized at the Montecatone Rehabilitation Institute. They are randomly assigned to Active tDCS (A) or Sham tDCS (S) (parallel arms design,1:1 allocation ratio). Two tDCS daily sessions for 5 days a week, for 2 consecutive weeks, are carried out simultaneously with the usual rehabilitation treatment of the upper limb, that is administered also at least 4 weeks before and 4 weeks after the tDCS treatment period.

Most outcomes are measured up to 4 weeks after the completion of the tDCS treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI;
* SCI neurological level, according to the American Spinal Injury Association (ASIA) definitions, from C3 to C7, included;
* incomplete SCI (i.e. ASIA Impairment Scale: B, C or D);
* distance from the SCI event: from 3 to 6 months;
* residual motor ability of the target upper limb;
* stable clinical conditions;
* tolerance to sitting position for at least 45 minutes;
* subjects capable and collaborating, able to give informed consent in person.

Exclusion Criteria:

* presence of implanted devices (e.g. pacemakers, intrathecal infusers, neurostimulators, hearing aids);
* positive history of brain lesions;
* presence of cerebral metallic implants (clips) or intracranial implants (e.g. ventriculoperitoneal shunt);
* history of epilepsy or previous state of epileptic disease;
* mechanical ventilation in place;
* history of psychotic disorders;
* history of severe neurodegenerative disease;
* concomitant pre-existing clinical conditions that may interfere with movements of the target arm or hand (e.g. severe osteoarthritis, joint injuries, plexus injuries, peripheral nerve injuries, partial amputations);
* use of antiepileptic drugs blocking Sodium o Calcium channels (e.g. Carbamazepine) or N-Methyl-D-Aspartate receptor antagonists (e.g. Dextromethorphan);
* history of drugs abuse;
* further contraindications to the use of TMS for PEMs elicitation (e.g. migraine with aura, permanent head / face tattoos);
* presence of brain tumor;
* pregnancy in progress.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in motor function, after the tDCS treatment period completion | Baseline 1 (initial visit); Baseline 2 (second visit, 2 weeks after Baseline 1); just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1)
  Motor function (i.e. muscle strength) of the target upper limb, determined according to the Medical Research Council /International Classification for the Surgery of the Tetraplegic Hand (MRC/ICSTH)

SECONDARY OUTCOMES:
Permanence of motor function, 4 weeks after the tDCS treatment period completion | Just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1)
  Motor function (i.e. muscle strength) of the target upper limb, determined according to the Medical Research Council /International Classification for the Surgery of the Tetraplegic Hand (MRC/ICSTH)
Change in strength, sensitivity and grip, up to 4 weeks after the tDCS treatment period completion | Baseline 1 (initial visit); Baseline 2 (second visit, 2 weeks after Baseline 1); just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1)
  Strength, sensitivity and grip of the target upper limb, determined according to the Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP)
Change in spasticity, up to 4 weeks after the tDCS treatment period completion | Baseline 1 (initial visit); Baseline 2 (second visit, 2 weeks after Baseline 1); just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1)
  Spasticity of the target upper limb, determined according to the Modified Ashworth Scale (MAS)
Change in motor function and muscle activity during rest activity, from the beginning of the tDCS treatment period until 4 weeks after its completion | just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1)
  Motor function and muscle activity during rest activity, determined through Neurographic assessment of the following muscles: deltoid, biceps, carpus extensor, thumb abductor brevis
Change in Motor Evoked Potentials, from the beginning of the tDCS treatment period until 4 weeks after its completion | just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1)
  Motor Evoked Potentials (PEMs), elicited by Transcranial Magnetic Stimulation (TMS), of the following muscles: deltoid, biceps, carpus extensor, thumb abductor brevis
Pain, up to 4 weeks after the tDCS treatment period completion | Baseline 1 (initial visit); Baseline 2 (2 weeks after Baseline 1); just before tDCS session n.1 (4 weeks after Baseline 1); just after tDCS session n.20 (6 weeks after Baseline 1); 4 weeks after tDCS session n.20 (10 weeks after Baseline 1
  Pain assessment in the target upper limb, determined according to the Numeric Rating Scale (NRS)
Safety of the tDCS treatment | During and after each tDCS session (from week 4 to week 6 after Baseline 1); in the 4 weeks after tDCS session n.20 (up to 10 weeks after Baseline 1)
  Incidence of adverse events related to the tDCS treatments
Tolerability of the tDCS treatment | Just after tDCS session n.20 (week 6 after Baseline 1)
  Subjective patient's perception of the fatigue of the treatments with tDCS associated with the usual rehabilitation physiotherapy treatment of the upper limb, evaluated through a short in-house developed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Olivi, MD, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided